CLINICAL TRIAL: NCT00656864
Title: Effects of Pioglitazone on the Regulation of Insulin Secretion in Patients With Type 2 Diabetes
Brief Title: Pioglitazone Incretin Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: Takeda (Industry)
Responsible Party: Richard Pratley, MD, University of Vermont College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 08-107; GCRC-962
Record Dates: First submitted 2008-04-07; First posted 2008-04-11 (Estimated); Last update posted 2011-02-02 (Estimated); Status verified 2010-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes; pioglitazone; GIP
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Pioglitazone arm
  Interventions: Drug: Pioglitazone
- 2 (Placebo Comparator): Placebo arm
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pioglitazone — Starting dose at 15 mg for two weeks, then titrated up to 45 mg in the subsequent 2 weeks.
  Other Names: Actos (brand name for pioglitazone)
  Arms: 1
Drug: Placebo — placebo
  Arms: 2

SUMMARY:
Incretin hormones are hormones produced by the gut in response to food intake. These hormones help the body to control the metabolism of glucose (sugar). In particular, two incretin hormones (GLP-1 and GIP) cause the pancreas to secrete more insulin in response to high blood glucose levels. This helps the body to metabolize the glucose more effectively, lowering blood sugar levels. GLP-1 and GIP do not work as well in patients with type 2 diabetes (T2DM) as in subjects who do not have diabetes. This study tests whether a medicine called pioglitazone (Actos), which is commonly used to treat T2DM, improves the ability of GIP to increase insulin secretion.

To address this question the investigators will recruit patients with T2DM whose diabetes is controlled with either diet and exercise or with metformin (another medicine commonly used to treat T2DM). Subjects will undergo measurement of body fat by DEXA scanning and a series of studies to characterize their metabolism. These studies include an oral glucose tolerance test (a test sometimes used to diagnose diabetes), a mixed-meal challenge (to measure how much GLP-1 and GIP are produced in response to a meal) and measurement of insulin secretion in response to glucose and GIP given through a vein. The investigators will also obtain small samples of fat (from just under the skin of the belly) using a needle to measure levels of the receptor for GIP. Subjects will then be randomly assigned to 12 weeks of treatment with either pioglitazone or matching placebo (an inactive tablet that does not contain medication). The dose of pioglitazone will be increased during the first 4 weeks to the maximum prescribed dose of 45 mg per day. Subjects will be seen every 2-4 weeks during the treatment phase of the study. After 12 weeks of treatment all studies performed at the beginning of the study will be repeated. The pioglitazone treatment will continue until the end of testing, approximately 4 weeks.

The results of this study may give us information about why glucose control deteriorates in T2DM. This information might also lead to new ways to prevent or treat T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes controlled with diet+exercise or metformin monotherapy
* HbA1c less than or equal to 7%
* Women will be non-fertile or practicing birth control

Exclusion Criteria:

* Acute or chronic medical conditions that would contraindicate participation
* Class III or IV heart failure
* Pregnant or nursing women
* Patients taking antidiabetic medications other than metformin, oral or chronic topical steroids, weight loss agents, antipsychotics, or other drugs that could affect insulin sensitivity or secretion.
* AST or ALT more than 2.5 times the upper limit of normal
* Active alcohol or drug abuse
* Weight greater than 300 pounds

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-05; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Change in incretin-mediated insulin secretion and receptor regulation of glucose-dependent insulinotropic peptide (GIP) in patients with type 2 diabetes. | 12 weeks per subject

SECONDARY OUTCOMES:
Change in active GIP in response to an oral glucose tolerance test and mixed meal challenge | 12 weeks
Change in active GLP-1 in response to the oral glucose tolerance test and the mixed meal challenge | 12 weeks
Change in glucose response during the oral glucose tolerance test and mixed meal challenge | 12 weeks
Change in insulin secretion during the oral glucose tolerance test and the mixed meal challenge | 12 weeks
Change in the acute insulin response to glucose, insulin sensitivity and the disposition index during the IV glucose tolerance test. | 12 weeks
Change in adipocyte GIP receptor mRNA expression levels. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Pratley, MD, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont, South Burlington, Vermont, United States

REFERENCES:
- [Derived] Nunez Lopez YO, Casu A, Kovacova Z, Petrilli AM, Sideleva O, Tharp WG, Pratley RE. Coordinated regulation of gene expression and microRNA changes in adipose tissue and circulating extracellular vesicles in response to pioglitazone treatment in humans with type 2 diabetes. Front Endocrinol (Lausanne). 2022 Aug 31;13:955593. doi: 10.3389/fendo.2022.955593. eCollection 2022. PMID 36120427
- [Derived] Tharp WG, Gupta D, Sideleva O, Deacon CF, Holst JJ, Elahi D, Pratley RE. Effects of Pioglitazone on Glucose-Dependent Insulinotropic Polypeptide-Mediated Insulin Secretion and Adipocyte Receptor Expression in Patients With Type 2 Diabetes. Diabetes. 2020 Feb;69(2):146-157. doi: 10.2337/db18-1163. Epub 2019 Nov 22. PMID 31757794
- [Derived] Kovacova Z, Tharp WG, Liu D, Wei W, Xie H, Collins S, Pratley RE. Adipose tissue natriuretic peptide receptor expression is related to insulin sensitivity in obesity and diabetes. Obesity (Silver Spring). 2016 Apr;24(4):820-8. doi: 10.1002/oby.21418. Epub 2016 Feb 17. PMID 26887289